CLINICAL TRIAL: NCT05678296
Title: Investigation of Effectiveness of Local Antibiotic Applications With Platelet Rich Fibrin on Third Molar Surgery Outcomes In Vivo and In Vitro
Brief Title: Investigation of Effectiveness of Local Antibiotic With Platelet Rich Fibrin on Third Molar Surgery Outcomes In Vivo
Status: Completed | Type: Observational
Sponsor: Ceren Melahat Donmezer (Other)
Responsible Party: Sponsor-Investigator, Ceren Melahat Donmezer, Principal Investigator, Oral and Maxillofacial Surgeon, Near East University, Turkey
Organization: Near East University, Turkey (Other)
Other Study IDs: 67-774-2019
Record Dates: First submitted 2022-12-28; First posted 2023-01-10 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Impacted Wisdom Tooth; Pain; Staphylococcus Aureus
Keywords: local antibiotic; comparison; platelets rich fibrin
MeSH Terms: conditions — Pain; Staphylococcal Infections | interventions — Diagnosis; Analgesics; Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- control group: platelet-rich fibrin placed into the socket of extracted tooth and no antibiotic is prescribed.
  Interventions: Diagnostic Test: Diagnosis; Drug: Analgesic; Procedure: traditional osteotomies; Biological: Platelet Rich Fibrin
- group 1: platelet-rich fibrin + 0.5 ml amoklavin I.V. 1.2 gr placed into the socket of the extracted tooth.
  Interventions: Diagnostic Test: Diagnosis; Drug: Analgesic; Procedure: traditional osteotomies; Biological: Platelet Rich Fibrin; Drug: Antibiotic
- group 2: platelet-rich fibrin + 0.5 ml Clin 600 mg/4 ml IM/IV, 0.5 ml placed into the socket of the extracted tooth.
  Interventions: Diagnostic Test: Diagnosis; Drug: Analgesic; Procedure: traditional osteotomies; Biological: Platelet Rich Fibrin; Drug: Antibiotic

INTERVENTIONS:
Diagnostic Test: Diagnosis — All of the patients withstand a radiological examination, including panoramic radiography, and all were handled by the same surgeon and assistant.
Drug: Analgesic — Analgesics are prescribed for the patients for all groups.
Procedure: traditional osteotomies — In all groups the flap incision was triangular in shape which avoids muscle involvement (Archer flap).
Biological: Platelet Rich Fibrin — Platelet rich fibrin (PRF), is an example and popular procedure for accelerate healing of soft and hard tissue because of the presence of various growth factors.a blood sample was taken without anticoagulant in 10 mL glass-coated plastic tubes that were immediately centrifuged (Elektro-mag M415P) at 3,000 rpm for 10 min (approximately 400 g) (13). The platelet-poor plasma that accumulated at the top of the tubes was discarded.PRF was dissected approximately 2 mm below its contact point with the red corpuscles situated beneath, to include any remaining platelets that may have localized below the junction between the PRF and red corpuscles.
Drug: Antibiotic — no systemic antibiotics are prescribed for the patients for all groups.
  Groups: group 1; group 2

SUMMARY:
The aim of this study was investigate the effectiveness of Local Antibiotic Applications With Platelet Rich Fibrin on Third Molar Surgery Outcomes In Vivo and In Vitro. The study included a total of 60 patients with impacted mandibular third molar. Patients were evaluated in 3 randomly separated groups. For the first and second group, Platelets Rich Fibrin+ local antibiotics were applied into the tooth socket. For the first group, amoxicillin was applied and for the second group, clindamycin was applied. There was a control group which only Platelets Rich Fibrin was applied into the socket. The outcome variables were pain, swelling, the number of analgesics taken, and trismus. These variables were also assessed based on first, second, third, and seventh days following the operation.

ELIGIBILITY:
Inclusion Criteria:

* patient with no systemic diseases, no current infection, no smoke, no pregnancy

Exclusion Criteria:

* no inflammation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The patients with no systemic diseases aged between 19-45
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-04-23 (Actual)

PRIMARY OUTCOMES:
visual analogue scale (VAS) | Day 1
  It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.
visual analogue scale (VAS) | Day 2
  It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.
visual analogue scale (VAS) | Day 3
  It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.
visual analogue scale (VAS) | Day 7
  It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.
visual analogue scale (VAS) | Day 15
  It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.
swelling | Day 1
  measured using a flexible plastic measuring tape as described by Gabka and Matsumura by measuring the distance from the corner of the mouth to the attachment of the earlobe following the bulge of the cheek and the distance from the outer canthus of the eye to the angle of the mandible.
swelling | Day 2
  measured using a flexible plastic measuring tape as described by Gabka and Matsumura by measuring the distance from the corner of the mouth to the attachment of the earlobe following the bulge of the cheek and the distance from the outer canthus of the eye to the angle of the mandible.
swelling | Day 3
  measured using a flexible plastic measuring tape as described by Gabka and Matsumura by measuring the distance from the corner of the mouth to the attachment of the earlobe following the bulge of the cheek and the distance from the outer canthus of the eye to the angle of the mandible.
swelling | Day 7
  measured using a flexible plastic measuring tape as described by Gabka and Matsumura by measuring the distance from the corner of the mouth to the attachment of the earlobe following the bulge of the cheek and the distance from the outer canthus of the eye to the angle of the mandible.
swelling | Day 15
  measured using a flexible plastic measuring tape as described by Gabka and Matsumura by measuring the distance from the corner of the mouth to the attachment of the earlobe following the bulge of the cheek and the distance from the outer canthus of the eye to the angle of the mandible.
Trismus | Day 1
  Trismus by measuring the distance between the mesial incisal corners of the upper and lower right incisors during maximum mouth opening.
Trismus | Day 2
  Trismus by measuring the distance between the mesial incisal corners of the upper and lower right incisors during maximum mouth opening.
Trismus | Day 3
  Trismus by measuring the distance between the mesial incisal corners of the upper and lower right incisors during maximum mouth opening.
Trismus | Day 7
  Trismus by measuring the distance between the mesial incisal corners of the upper and lower right incisors during maximum mouth opening.
Trismus | Day 15
  Trismus by measuring the distance between the mesial incisal corners of the upper and lower right incisors during maximum mouth opening.

OTHER OUTCOMES:
Amount of analgesic tablets | day 1,2,3,7 and 15
  Check the patients analgesic number of days 1,2,3,7 and 15.

CONTACTS AND LOCATIONS:
Overall Officials: Ceren Melahat Dönmezer, Principal Investigator — Near East University
Locations (1):
- Near east University, Nicosia, Lefkosa, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Donmezer CM, Bilginaylar K. Comparison of the Postoperative Effects of Local Antibiotic versus Systemic Antibiotic with the Use of Platelet-Rich Fibrin on Impacted Mandibular Third Molar Surgery: A Randomized Split-Mouth Study. Biomed Res Int. 2021 Dec 2;2021:3040661. doi: 10.1155/2021/3040661. eCollection 2021. PMID 34901267
- [Result] Caymaz MG, Uyanik LO. Comparison of the effect of advanced platelet-rich fibrin and leukocyte- and platelet-rich fibrin on outcomes after removal of impacted mandibular third molar: A randomized split-mouth study. Niger J Clin Pract. 2019 Apr;22(4):546-552. doi: 10.4103/njcp.njcp_473_18. PMID 30975961
- [Result] Polak D, Clemer-Shamai N, Shapira L. Incorporating antibiotics into platelet-rich fibrin: A novel antibiotics slow-release biological device. J Clin Periodontol. 2019 Feb;46(2):241-247. doi: 10.1111/jcpe.13063. PMID 30629300
- [Result] Uyanik LO, Bilginaylar K, Etikan I. Effects of platelet-rich fibrin and piezosurgery on impacted mandibular third molar surgery outcomes. Head Face Med. 2015 Jul 26;11:25. doi: 10.1186/s13005-015-0081-x. PMID 26209242